CLINICAL TRIAL: NCT00002360
Title: Pivotal Bioequivalence Study of Videx Chewable/Dispersible Buffered Tablets and an Encapsulated Enteric Coated Bead Formulation of Didanosine in HIV-Infected Subjects
Brief Title: A Study Comparing Two Forms of Didanosine in HIV-infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 039H; 31876; AI454-157
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Didanosine; Tablets; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Therapeutic Equivalency
MeSH Terms: conditions — HIV Infections | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if the coated-capsule form of didanosine (ddI) is as safe and absorbed by the body as well as the chewable-tablet form of ddI.

Didanosine (ddI) is an anti-HIV drug. The effectiveness of ddI can be lowered by acid in the stomach. To prevent this, patients take antacids with ddI. The coated-capsule form of ddI may replace the need for antacids.

DETAILED DESCRIPTION:
Didanosine, a purine nucleoside analogue, is indicated for the treatment of HIV infection when antiretroviral therapy is warranted. Didanosine is administered orally with antacids to protect it against acid-induced hydrolysis in the stomach. To eliminate the need for using buffers in the ddI formulations, an enteric-coated bead formulation of ddI is being developed.

Patients are randomized to 1 of 2 groups to receive treatment on 2 separate occasions at least 72 hours apart. Group 1 receives the reference formulation of ddI. Group 2 receives the test formulation of ddI. Clinical evaluations, including clinical laboratory tests, are performed periodically during the study and at discharge. Serial blood samples are collected at specific time points over the 12 hours following dosing, and are used for the pharmacokinetic variables CMAX and AUC(INF). Factors used in analysis are sequence, subject within sequence, period, and formulation. Safety is assessed by monitoring adverse effects, vital signs, ECG recordings, and clinical laboratory tests throughout the study.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 cell counts of at least 200 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Any evidence of organ dysfunction.
* Any clinically significant deviations from specified baseline requirements for physical examinations, laboratory tests, or 12-lead electrocardiogram.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 1999-03; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A. Knupp, Study Director